CLINICAL TRIAL: NCT06427798
Title: Phase I/II Trial of Systemic Targeted Radioligand Therapy (TRT) With Somatostatin-Receptors (SSTR)-Agonist [212Pb]VMT-alpha-NET in Metastatic or Inoperable SSTR Positive (SSTR+) Gastrointestinal (GI) Neuroendocrine Tumors (NET) and Pheochromocytoma/Paragangliomas Previously Treated With Systemic Radioligand Therapy
Brief Title: Somatostatin-Receptors (SSTR)-Agonist [212Pb]VMT-alpha-NET in Metastatic or Inoperable SSTR+ Gastrointestinal Neuroendocrine Tumor and Pheochromocytoma/Paraganglioma Previously Treated With Systemic Targeted Radioligand Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001711; 001711-C
Record Dates: First submitted 2024-05-23; First posted 2024-05-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11-21

CONDITIONS: Somatostatin Receptor Positive; Gastrointestinal Neuroendocrine Tumors; Pheochromocytoma; Paragangliomas
Keywords: 212Pb; Targeted Therapy; Image-Guided Dosimetry; VMT- -NET
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Dosimetry Arm 1 (Experimental): Escalating doses of [212Pb]VMT-alpha-NET, imaging with [203Pb]VMT-alpha-NET.
  Interventions: Drug: 68Ga-DOTATATE; Drug: [203Pb]VMT-alpha-NET; Drug: [212Pb]VMT-alpha-NET
- 2/Arm 2 (Experimental): Escalating doses of [212Pb]VMT-alpha-NET.
  Interventions: Drug: 68Ga-DOTATATE; Drug: [212Pb]VMT-alpha-NET
- 3/Arm 3 (Experimental): [212Pb]VMT-alpha-NET at MTD.
  Interventions: Drug: 68Ga-DOTATATE; Drug: [212Pb]VMT-alpha-NET

INTERVENTIONS:
Drug: 68Ga-DOTATATE — 68Ga-DOTATATE PET/CT whole-body scanning will be done at target dose of 5 mCi. The whole-body PET/CT scan will be started approximately 60 minutes after the tracer injection and will take up to 2 hours.
Drug: [203Pb]VMT-alpha-NET — [203Pb]VMT-alpha-NET (6 mCi) will be given IV at 7 days prior.
  Arms: 1/Dosimetry Arm 1
Drug: [212Pb]VMT-alpha-NET — [212Pb]VMT-alpha-NET will be given IV on Day 1 of every cycle for 4 cycles total at escalating doses in Phase I and at MTD during Phase II. One cycle is 8 weeks.

SUMMARY:
Background:

Gastrointestinal neuroendocrine tumors (GI NET) are a type of cancer that affects the stomach and intestines; pheochromocytoma/paragangliomas (PPGL) are tumors that grow in or near the adrenal glands. Both of these types of tumor have high levels of a protein called somatostatin receptors (SSTR) on their surfaces. Researchers want to test a treatment that targets SSTR.

Objective:

To test a drug ([212Pb]VMT-alpha-NET) in people with GI NET or PPGL. The drug has 2 components: a protein to bind to SSTR and a radioactive agent to kill the cancer cells.

Eligibility:

Adults aged 18 years or older with GI NET or PPGL tumors that have spread and cannot be removed with surgery.

Design:

Participants will be screened. They will have a physical exam, with imaging scans, blood tests, and tests of their heart function.

[212Pb]VMT-alpha-NET is given through a tube attached to a needle inserted into a vein (infusion). Treatment will be given in four 8 week cycles. Participants will receive the drug on the first day of each cycle. They will remain in the clinic at least 4 hours after each infusion and may need to stay in the hospital for up to 48 hour for monitoring and testing. They will have blood tests every week of each cycle.

Some participants will also get a related study drug ([203Pb]VMT-alpha-NET). They will receive this drug a few days before the first 2 cycles. At 4, 24, and 48 hours after each infusion, they will have whole body scans. These scans will show where the study drug went in their body.

Follow-up visits will continue for 10 years....

DETAILED DESCRIPTION:
Background:

* Somatostatin receptors (SSTR) have been shown to be over-expressed in a number of human tumors, including gastrointestinal (GI) neuroendocrine tumors (NET) and pheochromocytoma/paragangliomas (PPGL).
* Targeted radioligand therapy (TRT) is a class of cancer therapeutic agents formed by attaching a radioactive isotope to a ligand that can target specific surface receptors such as SSTR on a tumor cell membrane. Efficacy is typically determined by the radiation dose deposited onto a tumor, which is determined by the radioactive isotope being used as well as the binding characteristics of the ligand-receptor/transporter pair.
* While there have been clinical successes with treating gastrointestinal neuroendocrine tumors (GI NET) and PPGL with SSTR-targeting beta-emitting TRTs, tumors will invariably start to progress after some time. Re-treatment using the same beta-emitting agents at the time of progression can be done but has decreased efficacy compared to the TRT-naive setting.
* Alpha emitters such as 212Pb emit alpha particles that are more damaging to tumor cells than beta emitters such as 177Lu. Therefore, TRT agents using alpha emitters are considered to be more potent and could be better than betas in the re-treatment setting.
* VMT-alpha-NET is a peptide that binds to SSTR, which when attached to 212Pb becomes an alpha particle-emitting TRT that can be used to treat tumors that have SSTR surface expression.
* [203Pb]VMT-alpha-NET is the chemically identical imaging surrogate for [212Pb]VMT-alpha-NET and has the same mechanism of action via binding to SSTR2. The nuclide 203Pb contained in [203Pb]VMT-alpha-NET emits gamma radiation suitable for single-photon emission computerized tomography (SPECT) imaging. These images can be used to assess drug product biodistribution throughout the body.

Objectives:

* Phase I: To determine the maximal tolerated dose (MTD) of [212Pb]VMT-alpha-NET using a 3+3 dose escalation design in GI NET and PPGL in a re-treatment setting.
* Phase II: To determine the Overall Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of participants treated with [212Pb]VMT-alpha-NET at the MTD at the completion of 4 cycles of treatment, reported by disease groups.

Eligibility:

* Age >= 18 years.
* Histopathologically confirmed GI NET or PPGL that are metastatic or inoperable.
* At least 1 prior systemic radioligand therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status <= 1.

Design:

* This is an open-label, single-arm, single-center, phase I/II study evaluating the safety, preliminary efficacy, and pharmacokinetic properties of [212Pb]VMT-alpha-NET in GI NET and PPGL in a re-treatment setting.
* Phase I participants will be accrued using a 3+3 dose escalation design with 3 dose levels to estimate MTD of [212Pb]VMT-alpha-NET. Once MTD is estimated, Phase II participants with GI NET and PPGL will be accrued in separate cohorts and treated at MTD of [212Pb]VMT-alpha-NET.
* [212Pb]VMT-alpha-NET will be given IV every 8 weeks for a total of 4 administrations.
* A subset of participants (Dosimetry Arm 1) will have [203Pb]VMT-alpha-NET administration followed by whole-body gamma scans combined with dosimetry SPECT/ Computed Tomography (CT) scans and collection of blood and urine samples prior to each cycle.
* Participants will have timed clinical laboratory evaluations, imaging studies, and research blood, and urine samples while on the study therapy for safety and efficacy evaluations.
* Following completion of treatment, participants will be seen at the NIH Clinical Center approximately 30 days later, every 12 weeks for years 1-3, every 6 months for years 4-6 for safety and efficacy assessments. Beyond 6 years, participants will be contacted annually through any NIH-approved platform to assess for overall survival and health status.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histopathologically confirmed gastrointestinal neuroendocrine tumors (GI NET) or pheochromocytoma/paraganglioma (PPGL) cancers that are metastatic or inoperable per Standard of Care.
* Have received at least 1 prior systemic radioligand therapy for definitive therapeutic purposes. Note: Participants with prior external beam radiation treatment (EBRT) will also be eligible as long as they have had at least 1 prior administration of a systemic radioligand therapy.
* Must have at least 1 measurable lesion by RECIST 1.1 (phase II only).
* History of progression by imaging (e.g., RECIST 1.1) or clinically (defined as increase in severity or frequency of symptoms related to disease) within the past 36 months prior to the first dose of [203Pb]VMT-alpha-NET.
* Evidence of somatostatin receptors (SSTR) expression on at least 50 percent of the radiographically identifiable (i.e., visible on an anatomic scan such as CT or magnetic resonance imaging [MRI]) tumor, as indicated by a positive (uptake qualitatively identifiable as above the local background) on SSTR PET scan.
* Age >= 18 years.
* ECOG performance status <= 1.
* Participants must have adequate organ and marrow function as defined below:

  * Leukocytes: 3,000/microliter
  * Absolute Neutrophil Count: 1,500/microliter
  * Platelets: 100,000/miroliter
  * Hemoglobin: >= 9.0 g/dL
  * Total bilirubin: within normal institutional limits. Note: <= 5 X institutional upper limit of normal (ULN) if bilirubin elevation is due to a benign process such as Gilbert syndrome
  * AST: <= 2.5 X institutional ULN
  * ALT: <= 2.5 X institutional ULN
  * Creatinine: within normal institutional limits

OR

* Calculated creatinine clearance (glomerular filtration rate (eGFR): >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal

  * Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression at screening.
  * Participants with new or progressive brain metastases or leptomeningeal disease are eligible as long as the participant is asymptomatic and not requiring medication for symptom control from the brain lesions at screening.
  * Participants seropositive for human immunodeficiency virus (HIV) must:
* be on effective anti-retroviral therapy; and
* have an undetectable viral load at screening.
* Participants seropositive for hepatitis B virus (HBV), must have HBV viral load undetectable at screening.

  -Participants seropositive for hepatitis C virus (HCV) must:
* received curative treatment; and
* have an undetectable HCV viral load at screening.

  * Participants may enroll in this study while on another therapeutic trial in order to start the screening process. However, all other investigational agents should be stopped at least 28 days prior to receiving [203Pb]VMT-alpha-NET.
  * Individuals of child-bearing potential (IOCBP) and individuals who can father children must agree to use an effective method of contraception (barrier, hormonal, intrauterine device [IUD], surgical sterilization, abstinence) at study entry and at least 6 months after the last dose of the study agent(s).
  * Nursing participants must be willing to discontinue nursing from study treatment initiation through 6 months after the last dose of the study agents.
  * The ability of the participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to VMT-alpha-NET.
* Positive Beta human chorionic gonadotropin (Beta-HCG) serum or urine pregnancy test performed in i IOCBP at screening.
* QTc > 450 ms on electrocardiogram (EKG) at screening. Note: Framingham correction for QTc will be used
* History of or detection at screening of active/untreated secondary malignancy except nonmelanoma skin cancer and carcinoma in situ of the uterine cervix.
* Uncontrolled intercurrent illness, factors, evaluated by medical history and physical exam which would potentially increase in the risk of the participant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2039-07-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: MTD of [212Pb]VMT-alpha-NET using a 3+3 dose escalation design in GI NET and PPGL in a re-treatment setting | DLT period (through 12 weeks after initial 212Pb]VMT-alpha-NET administration).
  The MTD will be presented as a recommended dose to be used as the recommended phase II dose (RP2D) for the combined participant population, as well as for each disease group being studied (GI-NET, PPGL).
Phase II: ORR by RECIST 1.1 of participants treated with [212Pb]VMT-alpha-NET at the MTD at the completion of 4 cycles of treatment, reported by disease groups | Baseline until progression or 6 years after receiving the first infusion of study drug.
  The overall response rate will be presented as a percentage along with 95% confidence intervals. Only evaluable participants will be included.

SECONDARY OUTCOMES:
Progression Free Survival | Baseline until progression or 10 years after receiving the first infusion of study drug
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Kaplan-Meier curves of PFS will be constructed. Median PFS will be reported with 95% confidence intervals.
Safety of [203Pb]VMT-alpha-NET and [212Pb]VMT-alpha-NET | Study duration
  Descriptive tabulations of toxicity will be provided, along with the agent attribution determination and CTCAE grade for each toxicity event. The data will be presented as an absolute count of the event at a participant level as well as a percentage of total evaluable participants.
Overall Survival | Baseline until progression or 10 years after receiving the first infusion of study drug
  Kaplan-Meier curves of OS, will be constructed. Median OS will be reported with 95% confidence intervals.
PK properties of [212Pb]VMT-alpha-NET via blood and urine sampling | After every infusion of [212Pb]VMT-alpha-NET
  PK data will be represented as a scatter plot graphing time vs. the amount of radioactivity found in blood and urine samples.
Dosimetry properties of [212Pb]VMT-alpha-NET via SPECT/CT, using [203Pb]VMT-alpha-NET as a surrogate with and without the administration of amino acids (Dosimetry Arm 1 only) | In Dosimetry Arm 1 after every [203Pb]VMT-alpha-NET infusion
  Biodistribution and dosimetry data will be represented in a tabular format which indicates the percentage of the injected dose calculated to be in each of the major organs using gamma scan results. Radiation dose calculations will be performed using OLINDA/EXM software. Absorbed doses in organs and the whole body will be determined using the appropriate adult phantom (e.g., adult male, adult female). Tumor lesion absorbed doses will be determined using the sphere model in OLINDA.

CONTACTS AND LOCATIONS:
Overall Officials: Frank I Lin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested by other researchers after the completion of the primary endpoint.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001711-C.html